CLINICAL TRIAL: NCT03318094
Title: Vanderbilt University Medical Center
Brief Title: Role of Sympathetic Vasoconstriction on Insulin-Mediated Microvascular Recruitment and Glucose Uptake in Obesity
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Italo Biaggioni, Professor Medicine and Pharmacology, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 162097
Record Dates: First submitted 2017-10-17; First posted 2017-10-23 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Insulin Resistance; Healthy; Obesity
Keywords: insulin resistance; phentolamine; microvascular recruitment; autonomic nervous system
MeSH Terms: conditions — Insulin Resistance; Obesity | interventions — Phentolamine; Adrenergic alpha-Antagonists; Sodium Chloride; Nitroprusside

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intact Day (Placebo Comparator): Saline
  Interventions: Other: Saline
- Blocked Day (Experimental): Phentolamine
  Interventions: Drug: Phentolamine
- Vasodilator Comparison (Active Comparator): Sodium Nitroprusside
  Interventions: Drug: Sodium Nitroprusside

INTERVENTIONS:
Drug: Phentolamine — Intrabrachial phentolamine will be given on the blocked day
  Other Names: alpha-adrenergic blocker
  Arms: Blocked Day
Other: Saline — Intrabrachial saline will be given this day
  Arms: Intact Day
Drug: Sodium Nitroprusside — Intrabrachial sodium nitroprusside will be given this day to compare with phentolamine
  Other Names: Active comparison
  Arms: Vasodilator Comparison

SUMMARY:
The purpose of this study is to better understand the contribution of sympathetic vasoconstriction to impaired insulin-mediated vasodilation and subsequently insulin-mediated glucose uptake. The investigators will test the hypothesis that removal of sympathetic vasoconstriction can result in improvement in insulin-mediated vasodilation and subsequently sensitivity to insulin-mediated glucose uptake.

DETAILED DESCRIPTION:
Several studies have shown that obese subjects have impaired Nitric Oxide (NO)-mediated dilation; and those who develop insulin resistance tend to be more obese, have higher insulin levels and greater sympathetic activity. Furthermore, we have made the novel observation that autonomic blockade improves glucose utilization in obese subjects with insulin resistance, providing a causal relation between sympathetic activation and insulin resistance. The autonomic blockade also improved NO-mediated dilation in obese subjects, which may improve glucose uptake by promoting glucose delivery.

The investigators will enroll obese insulin-resistant subjects and in parallel experiments two comparator groups: obese insulin sensitive subjects, and healthy lean control subjects. We will assess the effects of insulin (hyperinsulinemic euglycemic clamp) on microvascular recruitment, and forearm glucose uptake on two separate occasions randomly assigned and at least one month apart, during an intrabrachial infusion of the alpha-adrenergic blocker phentolamine (blocked day) or saline control (Control day).

ELIGIBILITY:
Inclusion Criteria:

* Males and females of all races between 18 and 60 years of age.
* Obesity defined as body mass index between 30-40 kg/m2
* Insulin resistance defined as homeostasis model assessment 2 insulin resistance (HOMA2-IR) score >1.6 (never diagnosed or treated type 2 diabetic), or being a well-controlled type 2 diabetic on metformin only.
* Able and willing to provide informed consent

Exclusion Criteria:

* Pregnancy or breastfeeding
* Current smokers or history of heavy smoking (>2 packs/day)
* History of alcohol or drug abuse
* Morbid obesity (BMI > 40 kg/m2)
* Previous allergic reaction to study medications
* Evidence of type I diabetes.
* Cardiovascular disease other than hypertension such as myocardial infarction within 6 months prior to enrollment, presence of angina pectoris, significant arrhythmia, congestive heart failure (LV hypertrophy acceptable), deep vein thrombosis, pulmonary embolism, second or third-degree heart block, mitral valve stenosis, aortic stenosis, or hypertrophic cardiomyopathy
* History of serious cerebrovascular disease such as cerebral hemorrhage, stroke, or transient ischemic attack
* History or presence of immunological or hematological disorders
* Impaired hepatic function [aspartate amino transaminase (AST) and/or alanine amino transaminase (ALT) > 2.0 x upper limit of normal range]
* Impaired renal function (serum creatinine >1.5 mg/dl)
* Moderate to severe anemia (hemoglobin <11 g/dl)
* Treatment with serotonin-norepinephrine reuptake inhibitors (SNRIs) or norepinephrine transporter (NET) inhibitors
* Treatment with phosphodiesterase 5 inhibitors
* Treatment with anticoagulants
* Treatment with chronic systemic glucocorticoid therapy (more than 7 consecutive days in 1 month)
* Treatment with any investigational drug in the 1 month preceding the study
* Inability to give, or withdraw, informed consent
* Other factors which in the investigator's opinion would prevent the subject from completing the protocol (i.e., clinically significant abnormalities on clinical, mental examination or laboratory testing or inability to comply with protocol)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2017-10-24 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Contrast Enhanced-Ultrasonography (CEU) | Before clamp and 15 minutes after clamp
  The Primary Outcome will be the change in CEU induced by insulin during hyperinsulinemic clamp compared to baseline. To test the null hypothesis that insulin will not produce any changes in microvascular blood volume using CEU in response to α-adrenergic blockade (phentolamine) in the isolated forearm model.

CONTACTS AND LOCATIONS:
Locations (1):
- Autonomic Dysfunction Center, Nashville, Tennessee, United States